CLINICAL TRIAL: NCT00075725
Title: High Risk B-Precursor Acute Lymphoblastic Leukemia (ALL)
Brief Title: Dexamethasone Compared With Prednisone During Induction Therapy and Methotrexate With or Without Leucovorin During Maintenance Therapy in Treating Patients With Newly Diagnosed High-Risk Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AALL0232; NCI-2009-00301 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AALL0232; CDR0000349182; 11723; AALL0232 (Other: Children's Oncology Group); AALL0232 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Results first posted 2015-08-06 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Acute Lymphoblastic Leukemia; Adult B Acute Lymphoblastic Leukemia; Childhood B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Leucovorin; Mercaptopurine; azathiopurine; Methotrexate; merphos; pegaspargase; Prednisone; deltacortene; prednylidene; Radiotherapy; Radiation; Thioguanine; Vincristine

ARMS (4):
- Arm I (Active Comparator): Patients in arm I receive intrathecal cytarabine in week 1; infusions of vincristine and daunorubicin once a week in weeks 1-4; dexamethasone by mouth or infusion twice a day in weeks 1 and 2; intrathecal methotrexate in weeks 2 and 5 or 2-5; and an injection of pegaspargase in week 1.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Radiation: Radiation Therapy; Drug: Thioguanine; Drug: Vincristine Sulfate
- Arm II (Active Comparator): Patients in arm II will receive intrathecal cytarabine in week 1; infusions of vincristine and daunorubicin once a week in weeks 1-4; dexamethasone by mouth or infusion twice a day in weeks 1 and 2; intrathecal methotrexate in weeks 2 and 5 or 2-5; and an injection of pegaspargase in week 1.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Radiation: Radiation Therapy; Drug: Thioguanine; Drug: Vincristine Sulfate
- Arm III (Experimental): Patients in arm III will receive cytarabine, vincristine, daunorubicin, and pegaspargase as in groups one and two. They will also receive prednisone by mouth or infusion twice a day in weeks 1-4 and intrathecal methotrexate in weeks 2 and 5.
  Some patients in all groups may receive induction therapy for 2 additional weeks. Beginning in week 6 or 7, patients may receive combination chemotherapy by infusion, injection, intrathecally, and by mouth for up to 8 weeks.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisone; Radiation: Radiation Therapy; Drug: Thioguanine; Drug: Vincristine Sulfate
- Arm IV (Experimental): Patients in arm IV will receive cytarabine, vincristine, daunorubicin, and pegaspargase as in groups one and two. They will also receive prednisone by mouth or infusion twice a day in weeks 1-4 and intrathecal methotrexate in weeks 2 and 5.
  Some patients in all groups may receive induction therapy for 2 additional weeks. Beginning in week 6 or 7, patients may receive combination chemotherapy by infusion, injection, intrathecally, and by mouth for up to 8 weeks.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisone; Radiation: Radiation Therapy; Drug: Thioguanine; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IT, SC, or IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
  Arms: Arm II; Arm IV
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IT or IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Pegaspargase — Given IM
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Drug: Prednisone — Given PO or IV
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
  Arms: Arm III; Arm IV
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Thioguanine — Given PO
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This randomized phase III trial is studying dexamethasone to see how well it works compared to prednisone during induction therapy. This trial is also studying methotrexate and leucovorin calcium to see how well they work compared to methotrexate alone during maintenance therapy in treating patients with newly diagnosed acute lymphoblastic leukemia (ALL). Drugs used in chemotherapy, such as dexamethasone, prednisone, methotrexate, and leucovorin calcium, work in different ways to stop cancer cells from dividing so they stop growing or die. Giving more than one drug may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective in treating acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Improve the outcome of children with high-risk acute lymphoblastic leukemia treated with 2 different chemotherapy regimens.

II. Determine the relative safety and efficacy of dexamethasone given for 14 days vs prednisone given for 28 days during induction.

III. Determine the relative safety and efficacy of high-dose methotrexate (5gm/m^2) with leucovorin rescue compared to escalating methotrexate without leucovorin rescue (Capizzi I) during interim maintenance I.

IV. Correlate Day 29 minimal residual disease (MRD) with event-free survival (EFS) and overall survival (OS).

V. Correlate early marrow response status with day-29 MRD status. VI. Improve outcome by identifying additional high risk patients by Day 29 MRD for treatment with fully augmented Berlin-Frankfurt-Munster (BFM).

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to early response (slow early response [SER] vs rapid early response [RER]). Induction therapy: Patients are randomized to 1 of 4 treatment arms.

ARM I: Patients receive cytarabine intrathecally (IT) on day 1, vincristine intravenously (IV) and daunorubicin IV on days 1, 8, 15, and 22, dexamethasone orally (PO) or IV twice daily (BID) on days 1-14, methotrexate (MTX) IT on days 8 and 29* and pegaspargase intramuscularly (IM) once on day 4, 5, or 6.

NOTE: *Patients with CNS3 disease (WBC > 5/mL in cerebrospinal fluid and positive for blasts on cytospin) also receive MTX IT on days 15 and 22.

ARM II: Patients receive induction therapy as in Arm I.

ARM III: Patients receive cytarabine, vincristine, daunorubicin, and pegaspargase as in Arm I. Patients also receive prednisone PO or IV BID on days 1-28 and MTX IT on days 8 and 29.

ARM IV: Patients receive induction therapy as in Arm III.

Patients in all arms are evaluated at day 29 of induction therapy. Patients with M3 disease are removed from study. Patients with M1 disease and less than 1% minimal residual disease (MRD) proceed to consolidation therapy beginning on day 36. Patients with M2 disease OR with MI disease and at least 1% MRD receive extended induction therapy for 2 additional weeks. Patients with SER disease and MLL rearrangements are removed from the study but may be eligible for treatment on protocol COG-AALL0031.

Extended induction therapy: Patients continue to receive therapy on the arm to which they were originally randomized.

ARMS I and II: Patients receive dexamethasone PO or IV BID on days 1-14, vincristine IV on days 1 and 8, daunorubicin IV on day 1 and pegaspargase IM on day 4, 5, or 6 and are then reevaluated.

ARMS III and IV: Patients receive prednisone PO or IV BID on days 1-14, and vincristine, daunorubicin, and pegaspargase as in Arms I and II and are then reevaluated.

Patients on all arms who have M1 disease and less than 1% MRD after extended induction proceed to consolidation therapy and continue as SER patients. All other patients are removed from study.

Consolidation therapy: All patients receive cyclophosphamide IV over 30 minutes on days 1 and 29, cytarabine IV or subcutaneously (SC) on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine (MP) PO on days 1-14 and 29-42, vincristine IV on days 15, 22, 43, and 50; pegaspargase IM on days 15 and 43 and MTX* IT on days 1, 8, 15, and 22. Patients with testicular disease also receive radiotherapy to the testes.

NOTE: *Patients with CNS3 disease receive MTX on days 1 and 8 only.

Interim maintenance therapy I: Patients continue to receive treatment on the arm to which they were originally randomized.

ARM I: (escalating-dose MTX) Patients receive vincristine IV and escalating-dose MTX IV on days 1, 11, 21, 31, and 41, pegaspargase IM on days 2 and 22 and MTX IT on days 1 and 21.

ARM II: (high-dose MTX) Patients receive vincristine IV and high-dose methotrexate IV over 24 hours on days 1, 15, 29, and 43, MP PO on days 1-56 and IT MTX on days 1 and 29. Patients also receive leucovorin calcium IV every 6 hours for at least 3 doses, beginning 42 hours after start of each MTX infusion.

ARM III: (escalating-dose MTX) Patients receive interim maintenance I therapy as in Arm I.

ARM IV: (high-dose MTX) Patients receive interim maintenance I therapy as in Arm II.

DELAYED INTENSIFICATION THERAPY I: All patients receive vincristine IV on days 1, 8, 15, 43, and 50, dexamethasone PO or IV BID on days 1 to 21 for patients age 1 to 12 OR on days 1-7 and 15-21 for patients age 13 and over, doxorubicin IV on days 1, 8, and 15, pegaspargase IM on day 4, 5, or 6 AND day 43, cyclophosphamide IV over 30 minutes on day 29, cytarabine IV or SC on days 30-33 and 37-40, thioguanine PO on days 29-42 and MTX IT on days 1, 29, and 36.After delayed intensification I, SER patients proceed to interim maintenance II and delayed intensification II. RER patients proceed directly to maintenance.

INTERIM MAINTENANCE THERAPY II: All patients receive vincristine IV and MTX IV on days 1, 11, 21, 31, and 41, pegaspargase IM on days 2 and 22; and MTX IT on days 1 and 21. Patients then proceed to delayed intensification II.

DELAYED INTENSIFICATION THERAPY II: All patients receive therapy as in delayed intensification I, arm I. CNS3 patients also receive radiotherapy for 3-10 days, beginning on day 29. All other SER patients, patients with MLL rearrangements, and some patients pretreated with steroids (> 48 hours within the week prior to diagnosis) receive prophylactic cranial radiotherapy (CRT) for 8 days, beginning on day 29. Patients then proceed to maintenance therapy.

MAINTENANCE THERAPY: All patients receive vincristine IV on days 1, 29, and 57, dexamethasone PO BID on days 1-5, 29-33, and 57-61, MP PO on days 1-84, MTX IT on day 1*; and MTX PO on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.

NOTE: *RER (who did not undergo CRT) patients also receive MTX IT on day 29 for maintenance courses 1-4.

In all arms, maintenance therapy repeats every 12 weeks until total duration of therapy is 2 years from the start of interim maintenance I for female patients and 3 years from the start of interim maintenance I for male patients. Patients with testicular disease may receive testicular radiotherapy for 8 days during one of the first 3 courses of maintenance therapy. Patients are followed monthly for 1 year, every 2 months for 1 year, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Must be eligible for and enrolled on classification study COG-AALL03B1
* Newly diagnosed B-precursor acute lymphoblastic leukemia

  * WBC > 50,000/mm^3 for patients age 1 to 9
  * Any WBC for patients age 10 to 30 OR patients who have received prior steroid therapy OR patients with testicular disease
* Whit blood cell (WBC) criteria:

  * Age 1 - 9 years: WBC >= 50,000/uL
  * Age 10 - 30 years: any WBC
  * Prior steroid therapy: any WBC
  * Testicular disease: any WBC
* Patients shall have had no other prior cytotoxic chemotherapy with the exception of steroids and intrathecal cytarabine
* Patients receiving prior steroid therapy (as described in AALL03B1) are eligible for study; the dose and duration of previous steroid therapy should be carefully documented
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with Down syndrome are ineligible to enroll onto this study

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3154 (Actual)
Dates: Start 2003-12-29 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Larsen, Principal Investigator — Children's Oncology Group
Locations (234):
- United States (208):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Beaumont Children's Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Children's Hospital and Clinic-Saint Paul, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Brookdale Hospital Medical Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Winthrop Hospital, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Oncology Group, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Victoria Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- New Zealand (3):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
  - Wellington Children's Hospital, Wellington
- Switzerland (3):
  - Swiss Pediatric Oncology Group - Bern, Bern
  - Swiss Pediatric Oncology Group - Geneva, Geneva
  - Swiss Pediatric Oncology Group - Lausanne, Lausanne

REFERENCES:
- [Derived] Chang TC, Chen W, Qu C, Cheng Z, Hedges D, Elsayed A, Pounds SB, Shago M, Rabin KR, Raetz EA, Devidas M, Cheng C, Angiolillo A, Baviskar P, Borowitz M, Burke MJ, Carroll A, Carroll WL, Chen IM, Harvey R, Heerema N, Iacobucci I, Wang JR, Jeha S, Larsen E, Mattano L, Maloney K, Pui CH, Ramirez NC, Salzer W, Willman C, Winick N, Wood B, Hunger SP, Wu G, Mullighan CG, Loh ML. Genomic Determinants of Outcome in Acute Lymphoblastic Leukemia. J Clin Oncol. 2024 Oct 10;42(29):3491-3503. doi: 10.1200/JCO.23.02238. Epub 2024 Aug 9. PMID 39121442
- [Derived] Escherich CS, Chen W, Li Y, Yang W, Nishii R, Li Z, Raetz EA, Devidas M, Wu G, Nichols KE, Inaba H, Pui CH, Jeha S, Camitta BM, Larsen E, Hunger SP, Loh ML, Yang JJ. Germ line genetic NBN variation and predisposition to B-cell acute lymphoblastic leukemia in children. Blood. 2024 May 30;143(22):2270-2283. doi: 10.1182/blood.2023023336. PMID 38446568
- [Derived] Rabin KR, Devidas M, Chen Z, Ji L, Kairalla J, Hitzler JK, Yang JJ, Carroll AJ, Heerema NA, Borowitz MJ, Wood BL, Roberts KG, Mullighan CG, Harvey RC, Chen IM, Willman CL, Reshmi SC, Gastier-Foster JM, Bhojwani D, Rheingold SR, Maloney KW, Mattano LA, Larsen EC, Schore RJ, Burke MJ, Salzer WL, Winick NJ, Carroll WL, Raetz EA, Loh ML, Hunger SP, Angiolillo AL. Outcomes in Children, Adolescents, and Young Adults With Down Syndrome and ALL: A Report From the Children's Oncology Group. J Clin Oncol. 2024 Jan 10;42(2):218-227. doi: 10.1200/JCO.23.00389. Epub 2023 Oct 27. PMID 37890117
- [Derived] Advani AS, Larsen E, Laumann K, Luger SM, Liedtke M, Devidas M, Chen Z, Yin J, Foster MC, Claxton D, Coffan K, Tallman MS, Appelbaum FR, Erba H, Stone RM, Hunger SP, McNeer JL, Loh ML, Raetz E, Winick N, Carroll W, Larson RA, Stock W. Comparison of CALGB 10403 (Alliance) and COG AALL0232 toxicity results in young adults with acute lymphoblastic leukemia. Blood Adv. 2021 Jan 26;5(2):504-512. doi: 10.1182/bloodadvances.2020002439. PMID 33496745
- [Derived] Wood B, Wu D, Crossley B, Dai Y, Williamson D, Gawad C, Borowitz MJ, Devidas M, Maloney KW, Larsen E, Winick N, Raetz E, Carroll WL, Hunger SP, Loh ML, Robins H, Kirsch I. Measurable residual disease detection by high-throughput sequencing improves risk stratification for pediatric B-ALL. Blood. 2018 Mar 22;131(12):1350-1359. doi: 10.1182/blood-2017-09-806521. Epub 2017 Dec 28. PMID 29284596
- [Derived] Karol SE, Mattano LA Jr, Yang W, Maloney KW, Smith C, Liu C, Ramsey LB, Fernandez CA, Chang TY, Neale G, Cheng C, Mardis E, Fulton R, Scheet P, San Lucas FA, Larsen EC, Loh ML, Raetz EA, Hunger SP, Devidas M, Relling MV. Genetic risk factors for the development of osteonecrosis in children under age 10 treated for acute lymphoblastic leukemia. Blood. 2016 Feb 4;127(5):558-64. doi: 10.1182/blood-2015-10-673848. Epub 2015 Nov 20. PMID 26590194
- [Derived] Karol SE, Yang W, Van Driest SL, Chang TY, Kaste S, Bowton E, Basford M, Bastarache L, Roden DM, Denny JC, Larsen E, Winick N, Carroll WL, Cheng C, Pei D, Fernandez CA, Liu C, Smith C, Loh ML, Raetz EA, Hunger SP, Scheet P, Jeha S, Pui CH, Evans WE, Devidas M, Mattano LA Jr, Relling MV. Genetics of glucocorticoid-associated osteonecrosis in children with acute lymphoblastic leukemia. Blood. 2015 Oct 8;126(15):1770-6. doi: 10.1182/blood-2015-05-643601. Epub 2015 Aug 11. PMID 26265699
- [Derived] Borowitz MJ, Wood BL, Devidas M, Loh ML, Raetz EA, Salzer WL, Nachman JB, Carroll AJ, Heerema NA, Gastier-Foster JM, Willman CL, Dai Y, Winick NJ, Hunger SP, Carroll WL, Larsen E. Prognostic significance of minimal residual disease in high risk B-ALL: a report from Children's Oncology Group study AALL0232. Blood. 2015 Aug 20;126(8):964-71. doi: 10.1182/blood-2015-03-633685. Epub 2015 Jun 29. PMID 26124497
- [Derived] Fernandez CA, Smith C, Yang W, Date M, Bashford D, Larsen E, Bowman WP, Liu C, Ramsey LB, Chang T, Turner V, Loh ML, Raetz EA, Winick NJ, Hunger SP, Carroll WL, Onengut-Gumuscu S, Chen WM, Concannon P, Rich SS, Scheet P, Jeha S, Pui CH, Evans WE, Devidas M, Relling MV. HLA-DRB1*07:01 is associated with a higher risk of asparaginase allergies. Blood. 2014 Aug 21;124(8):1266-76. doi: 10.1182/blood-2014-03-563742. Epub 2014 Jun 26. PMID 24970932

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexamethasone and Capizzi Methotrexate Patients < 10 Years; Dexamethasone & Capizzi Methotrexate Patients => 10 Years Old; Dexamethasone, Capizzi Methotrexate Down Syndrome (Non Random): Patients receive intrathecal cytarabine (Age-based dosing: Age (yrs) Dose 1 - 1.99 30 mg 2 - 2.99 50 mg ≥ 3 70 mg) on day 1; infusions of vincristine sulfate 1.5 mg/m2/dose (maximum dose of 2 mg) on Days 1, 8, 15 and 22 and daunorubicin hydrochloride (25 mg/m2/dose on Days 1, 8, 15 and 22. Dexamethasone (5 mg/m2/dose on Days 1-14 by mouth or infusion twice a day in weeks 1 and 2; intrathecal methotrexate (Aged based dosing: Age (yrs) Dose 1 - 1.99 8 mg 2 - 2.99 10 mg 3 - 8.99 12 mg ≥ 9 15 mg) on days 8 and 29 (CNS3 also on days 15 & 22) and an injection of pegaspargase (2500 International units/m2 x 1 dose on Day 4, 5 or 6).
- Dexamethasone, High Dose Methotrexate (Non Randomly Assigned): Patients non-randomly assigned to the DH (High Dose) regimen based on one (or more) of the following characteristics: (1) CNS3 status at entry, (2) testicular leukemic involvement at entry, or (3) extensive pre-treatment with steroids prior to entry. Patients receive intrathecal cytarabine (Age-based dosing: Age (yrs) Dose 1 - 1.99 30 mg 2 - 2.99 50 mg ≥ 3 70 mg) on day 1; infusions of vincristine sulfate 1.5 mg/m2/dose (maximum dose of 2 mg) on Days 1, 8, 15 and 22 and daunorubicin hydrochloride (25 mg/m2/dose on Days 1, 8, 15 and 22. Dexamethasone (5 mg/m2/dose on Days 1-14 by mouth or infusion twice a day in weeks 1 and 2; intrathecal methotrexate (Aged based dosing: Age (yrs) Dose 1 - 1.99 8 mg 2 - 2.99 10 mg 3 - 8.99 12 mg ≥ 9 15 mg) on days 8 and 29 (CNS3 also on days 15 & 22) and an injection of pegaspargase (2500 International units/m2 x 1 dose on Day 4, 5 or 6).
- Dexamethasone, High Dose Methotrexate (IM) < 10 Years; Dexamethasone, High Dose Methotrexate (IM) >= 10 Years: Patients randomly assigned to the DH regimen based on one (or more) of the following characteristics: (1) No CNS3 status at entry, (2) no testicular leukemic involvement at entry, or (3) no extensive pre-treatment with steroids prior to entry. Patients receive intrathecal cytarabine (Age-based dosing: Age (yrs) Dose 1 - 1.99 30 mg 2 - 2.99 50 mg ≥ 3 70 mg) on day 1; infusions of vincristine sulfate 1.5 mg/m2/dose (maximum dose of 2 mg) on Days 1, 8, 15 and 22 and daunorubicin hydrochloride (25 mg/m2/dose on Days 1, 8, 15 and 22. Dexamethasone (5 mg/m2/dose on Days 1-14 by mouth or infusion twice a day in weeks 1 and 2; intrathecal methotrexate (Aged based dosing: Age (yrs) Dose 1 - 1.99 8 mg 2 - 2.99 10 mg 3 - 8.99 12 mg ≥ 9 15 mg) on days 8 and 29 (CNS3 also on days 15 & 22) and an injection of pegaspargase (2500 International units/m2 x 1 dose on Day 4, 5 or 6).
- Prednisone, Capizzi Methotrexate <10 Years: Patients in regimen PC (Prednisone, Capizzi) will receive cytarabine, vincristine sulfate, daunorubicin hydrochloride, and pegaspargase. They will also receive prednisone by mouth or infusion twice a day in weeks 1-4 and intrathecal methotrexate in weeks 2 and 5. Some patients in all groups may receive induction therapy for 2 additional weeks. Beginning in week 6 or 7, patients may receive combination chemotherapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, mercaptopurine, cytarabine, thioguanine) by infusion, injection, intrathecally, and by mouth for up to 8 weeks.
- Prednisone, Capezzi Methotrexate >= 10 Years; Prednisone, Capezzi Methotrexate (Down's Syndrome): Patients in regimen PC will receive cytarabine, vincristine sulfate, daunorubicin hydrochloride, and pegaspargase. They will also receive prednisone by mouth or infusion twice a day in weeks 1-4 and intrathecal methotrexate in weeks 2 and 5. Some patients in all groups may receive induction therapy for 2 additional weeks. Beginning in week 6 or 7, patients may receive combination chemotherapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, mercaptopurine, cytarabine, thioguanine) by infusion, injection, intrathecally, and by mouth for up to 8 weeks.
- Prednisone and High Dose Methotrexate < 10 Yrs Old: Patients randomly assigned to the PH (Prednisone, High Dose MTX) regimen receive intrathecal cytarabine (Age-based dosing: Age (yrs) Dose 1 - 1.99 30 mg 2 - 2.99 50 mg ≥ 3 70 mg) on day 1; infusions of vincristine sulfate 1.5 mg/m2/dose (maximum dose of 2 mg) on Days 1, 8, 15 and 22 and daunorubicin hydrochloride (25 mg/m2/dose on Days 1, 8, 15 and 22. They will also receive prednisone by mouth or infusion twice a day in weeks 1-4 and intrathecal methotrexate in weeks 2 and 5. Some patients in all groups may receive induction therapy for 2 additional weeks. Beginning in week 6 or 7, patients may receive combination chemotherapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, mercaptopurine, cytarabine, thioguanine) by infusion, injection, intrathecally, and by mouth for up to 8 weeks.
- Prednisone and High Dose Methotrexate >=10 Years: Patients randomly assigned to the PH regimen receive intrathecal cytarabine (Age-based dosing: Age (yrs) Dose 1 - 1.99 30 mg 2 - 2.99 50 mg ≥ 3 70 mg) on day 1; infusions of vincristine sulfate 1.5 mg/m2/dose (maximum dose of 2 mg) on Days 1, 8, 15 and 22 and daunorubicin hydrochloride (25 mg/m2/dose on Days 1, 8, 15 and 22. They will also receive prednisone by mouth or infusion twice a day in weeks 1-4 and intrathecal methotrexate in weeks 2 and 5. Some patients in all groups may receive induction therapy for 2 additional weeks. Beginning in week 6 or 7, patients may receive combination chemotherapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, mercaptopurine, cytarabine, thioguanine) by infusion, injection, intrathecally, and by mouth for up to 8 weeks.
- Prednisone and High Dose Methotrexate (Non Randomly Assigned): Patients non-randomly assigned to the PH regimen based on one (or more) of the following: (1) CNS3 status at entry, (2) testicular leukemic involvement at entry, or (3) extensive pre-treatment with steroids prior to entry. Patients receive intrathecal cytarabine (Age-based dosing: Age (yrs) Dose 1 - 1.99 30 mg 2 - 2.99 50 mg ≥ 3 70 mg) on day 1; infusions of vincristine sulfate 1.5 mg/m2/dose (maximum dose of 2 mg) on Days 1, 8, 15 and 22 and daunorubicin hydrochloride (25 mg/m2/dose on Days 1, 8, 15 and 22. They will also receive prednisone by mouth or infusion twice a day in weeks 1-4 and intrathecal MTX in weeks 2 and 5. Some patients in all groups may receive induction therapy for 2 additional weeks. Beginning in week 6 or 7, patients may receive combination chemotherapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, mercaptopurine, cytarabine, thioguanine) by infusion, injection, intrathecally, and by mouth for up to 8 weeks.
Period: Overall Study
Arm/Group | Dexamethasone and Capizzi Methotrexate Patients < 10 Years | Dexamethasone, High Dose Methotrexate (Non Randomly Assigned) | Dexamethasone & Capizzi Methotrexate Patients => 10 Years Old | Dexamethasone, High Dose Methotrexate (IM) < 10 Years | Prednisone, Capizzi Methotrexate <10 Years | Prednisone, Capezzi Methotrexate >= 10 Years | Prednisone and High Dose Methotrexate < 10 Yrs Old | Prednisone and High Dose Methotrexate >=10 Years | Dexamethasone, High Dose Methotrexate (IM) >= 10 Years | Prednisone, Capezzi Methotrexate (Down's Syndrome) | Dexamethasone, Capizzi Methotrexate Down Syndrome (Non Random) | Prednisone and High Dose Methotrexate (Non Randomly Assigned)
Started | 246 | 106 | 296 | 246 | 232 | 710 | 246 | 696 | 302 | 34 | 12 | 28
Completed | 172 | 57 | 175 | 168 | 166 | 397 | 171 | 401 | 185 | 16 | 3 | 10
Not Completed | 74 | 49 | 121 | 78 | 66 | 313 | 75 | 295 | 117 | 18 | 9 | 18
Not completed — Adverse Event | 6 | 6 | 20 | 8 | 4 | 38 | 3 | 51 | 15 | 4 | 2 | 2
Not completed — Death | 3 | 5 | 10 | 2 | 3 | 25 | 4 | 22 | 14 | 4 | 3 | 0
Not completed — Lost to Follow-up | 1 | 1 | 4 | 1 | 0 | 13 | 2 | 4 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 6 | 5 | 8 | 4 | 19 | 3 | 17 | 5 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 3 | 3 | 2 | 1 | 2 | 3 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 12 | 3 | 6 | 10 | 6 | 27 | 7 | 31 | 10 | 2 | 0 | 0
Not completed — Disease Progression, all other reasons | 17 | 5 | 33 | 6 | 21 | 59 | 20 | 46 | 21 | 4 | 0 | 5
Not completed — Patient off treatment | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Ineligible or wrong diagnosis | 8 | 3 | 3 | 10 | 3 | 17 | 6 | 9 | 10 | 1 | 2 | 4
Not completed — Pt/Guardian refused RT therapy | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pt non compliant with therapy | 2 | 1 | 1 | 0 | 2 | 14 | 2 | 5 | 3 | 0 | 0 | 0
Not completed — Pt age out of range for treatment | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Insurance issues | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — MRD positive after extended ind | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Pt has very high risk ALL characteristic | 15 | 11 | 26 | 18 | 11 | 75 | 23 | 74 | 29 | 1 | 0 | 3
Not completed — Inevaluable | 1 | 1 | 4 | 2 | 2 | 9 | 1 | 11 | 2 | 0 | 1 | 0
Not completed — Other | 4 | 2 | 1 | 1 | 1 | 4 | 2 | 9 | 2 | 1 | 0 | 3
Not completed — Pt trying to find a BM donor | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Clinic chart lost unable to recreate | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unsuccessful institutional transfer | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — specimen(s) not submitted | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pt went to transplant | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pt received additional steroids | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pt relocated | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Institution Terminated | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Study Closure | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other complications | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pt care terminated due to pt behavior | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Pt incarcerated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dexamethasone, High Dose Methotrexate (Non Randomly Assigned): Patients non-randomly assigned to the DH regimen based on one (or more) of the following characteristics: (1) CNS3 status at entry, (2) testicular leukemic involvement at entry, or (3) extensive pre-treatment with steroids prior to entry. Patients receive intrathecal cytarabine (Age-based dosing: Age (yrs) Dose 1 - 1.99 30 mg 2 - 2.99 50 mg ≥ 3 70 mg) on day 1; infusions of vincristine sulfate 1.5 mg/m2/dose (maximum dose of 2 mg) on Days 1, 8, 15 and 22 and daunorubicin hydrochloride (25 mg/m2/dose on Days 1, 8, 15 and 22. Dexamethasone (5 mg/m2/dose on Days 1-14 by mouth or infusion twice a day in weeks 1 and 2; intrathecal methotrexate (Aged based dosing: Age (yrs) Dose 1 - 1.99 8 mg 2 - 2.99 10 mg 3 - 8.99 12 mg ≥ 9 15 mg) on days 8 and 29 (CNS3 also on days 15 & 22) and an injection of pegaspargase (2500 International units/m2 x 1 dose on Day 4, 5 or 6).
- Prednisone, Capizzi Methotrexate <10 Years; Prednisone, Capezzi Methotrexate >= 10 Years; Prednisone, Capezzi Methotrexate (Down's Syndrome): Patients in regimen PC will receive cytarabine, vincristine sulfate, daunorubicin hydrochloride, and pegaspargase. They will also receive prednisone by mouth or infusion twice a day in weeks 1-4 and intrathecal methotrexate in weeks 2 and 5. Some patients in all groups may receive induction therapy for 2 additional weeks. Beginning in week 6 or 7, patients may receive combination chemotherapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, mercaptopurine, cytarabine, thioguanine) by infusion, injection, intrathecally, and by mouth for up to 8 weeks.
- Prednisone and High Dose Methotrexate < 10 Yrs Old; Prednisone and High Dose Methotrexate >=10 Years: Patients randomly assigned to the PH regimen receive intrathecal cytarabine (Age-based dosing: Age (yrs) Dose 1 - 1.99 30 mg 2 - 2.99 50 mg ≥ 3 70 mg) on day 1; infusions of vincristine sulfate 1.5 mg/m2/dose (maximum dose of 2 mg) on Days 1, 8, 15 and 22 and daunorubicin hydrochloride (25 mg/m2/dose on Days 1, 8, 15 and 22. They will also receive prednisone by mouth or infusion twice a day in weeks 1-4 and intrathecal methotrexate in weeks 2 and 5. Some patients in all groups may receive induction therapy for 2 additional weeks. Beginning in week 6 or 7, patients may receive combination chemotherapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, mercaptopurine, cytarabine, thioguanine) by infusion, injection, intrathecally, and by mouth for up to 8 weeks.
- Dexamethasone, Capizzi Methotrexate Down Syndrome: Patients receive intrathecal cytarabine (Age-based dosing: Age (yrs) Dose 1 - 1.99 30 mg 2 - 2.99 50 mg ≥ 3 70 mg) on day 1; infusions of vincristine sulfate 1.5 mg/m2/dose (maximum dose of 2 mg) on Days 1, 8, 15 and 22 and daunorubicin hydrochloride (25 mg/m2/dose on Days 1, 8, 15 and 22. Dexamethasone (5 mg/m2/dose on Days 1-14 by mouth or infusion twice a day in weeks 1 and 2; intrathecal methotrexate (Aged based dosing: Age (yrs) Dose 1 - 1.99 8 mg 2 - 2.99 10 mg 3 - 8.99 12 mg ≥ 9 15 mg) on days 8 and 29 (CNS3 also on days 15 & 22) and an injection of pegaspargase (2500 International units/m2 x 1 dose on Day 4, 5 or 6).
- Prednisone and High Dose Methotrexate (Non Randomly Assigned): Patients non-randomly assigned to the PH regimen based on one (or more) of the following characteristics: (1) CNS3 status at entry, (2) testicular leukemic involvement at entry, or (3) extensive pre-treatment with steroids prior to entry. Patients receive intrathecal cytarabine (Age-based dosing: Age (yrs) Dose 1 - 1.99 30 mg 2 - 2.99 50 mg ≥ 3 70 mg) on day 1; infusions of vincristine sulfate 1.5 mg/m2/dose (maximum dose of 2 mg) on Days 1, 8, 15 and 22 and daunorubicin hydrochloride (25 mg/m2/dose on Days 1, 8, 15 and 22. They will also receive prednisone by mouth or infusion twice a day in weeks 1-4 and intrathecal methotrexate in weeks 2 and 5. Some patients in all groups may receive induction therapy for 2 additional weeks. Beginning in week 6 or 7, patients may receive combination chemotherapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, mercaptopurine, cytarabine, thioguanine) by infusion, injection, intrathecally, and by mouth
- Total: Total of all reporting groups
Arm/Group | Dexamethasone and Capizzi Methotrexate Patients < 10 Years | Dexamethasone, High Dose Methotrexate (Non Randomly Assigned) | Dexamethasone & Capizzi Methotrexate Patients => 10 Years Old | Dexamethasone, High Dose Methotrexate (IM) < 10 Years | Prednisone, Capizzi Methotrexate <10 Years | Prednisone, Capezzi Methotrexate >= 10 Years | Prednisone and High Dose Methotrexate < 10 Yrs Old | Prednisone and High Dose Methotrexate >=10 Years | Dexamethasone, High Dose Methotrexate (IM) >= 10 Years | Prednisone, Capezzi Methotrexate (Down's Syndrome) | Dexamethasone, Capizzi Methotrexate Down Syndrome | Prednisone and High Dose Methotrexate (Non Randomly Assigned) | Total
Number analyzed (Participants) | 246 | 106 | 296 | 246 | 232 | 710 | 246 | 696 | 302 | 34 | 12 | 28 | 3154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 246 | 96 | 275 | 246 | 232 | 641 | 246 | 610 | 266 | 30 | 10 | 26 | 2924
  Between 18 and 65 years | 0 | 10 | 21 | 0 | 0 | 69 | 0 | 86 | 36 | 4 | 2 | 2 | 230
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.0 (2.3) | 9.3 (6.0) | 14.1 (2.8) | 4.1 (2.2) | 4.2 (2.2) | 14.7 (3.3) | 4.2 (2.2) | 14.5 (3.2) | 14.6 (2.9) | 10.5 (5.7) | 12.3 (6.6) | 14.4 (2.9) | 10.8 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 31 | 135 | 117 | 106 | 321 | 108 | 288 | 128 | 18 | 7 | 11 | 1399
  Male | 117 | 75 | 161 | 129 | 126 | 389 | 138 | 408 | 174 | 16 | 5 | 17 | 1755
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 22 | 62 | 55 | 62 | 167 | 61 | 168 | 69 | 6 | 0 | 7 | 733
  Not Hispanic or Latino | 179 | 81 | 217 | 182 | 165 | 516 | 179 | 504 | 219 | 27 | 10 | 20 | 2299
  Unknown or Not Reported | 13 | 3 | 17 | 9 | 5 | 27 | 6 | 24 | 14 | 1 | 2 | 1 | 122
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 7 | 2 | 1 | 2 | 0 | 18
  Asian | 8 | 6 | 11 | 9 | 7 | 21 | 8 | 27 | 18 | 2 | 0 | 0 | 117
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 1 | 2 | 1 | 5 | 5 | 6 | 2 | 0 | 0 | 0 | 25
  Black or African American | 12 | 14 | 24 | 12 | 15 | 55 | 14 | 51 | 19 | 2 | 0 | 1 | 219
  White | 196 | 76 | 235 | 187 | 175 | 534 | 187 | 519 | 227 | 26 | 9 | 24 | 2395
  More than one race | 3 | 3 | 1 | 8 | 5 | 8 | 5 | 4 | 3 | 0 | 0 | 0 | 40
  Unknown or Not Reported | 25 | 6 | 24 | 27 | 29 | 83 | 26 | 82 | 31 | 3 | 1 | 3 | 340

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Increase in Cure Rate of High Risk ALL Without Causing More Serious Side Effects Between Interventions
Description: Event Free Probability.
Time Frame: 5 years
Population: Group "Prednisone and High Dose MTX (non-random)" who either had EFS events occur before 5 years or did not have minimum 5 years of follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Predisone and High Dose Methotrexate < 10 Yrs Old; Prenisone and High Dose Methotrexate >=10 Years: Patients randomly assigned to the PH regimen receive intrathecal cytarabine (Age-based dosing: Age (yrs) Dose 1 - 1.99 30 mg 2 - 2.99 50 mg ≥ 3 70 mg) on day 1; infusions of vincristine sulfate 1.5 mg/m2/dose (maximum dose of 2 mg) on Days 1, 8, 15 and 22 and daunorubicin hydrochloride (25 mg/m2/dose on Days 1, 8, 15 and 22. They will also receive prednisone by mouth or infusion twice a day in weeks 1-4 and intrathecal methotrexate in weeks 2 and 5. Some patients in all groups may receive induction therapy for 2 additional weeks. Beginning in week 6 or 7, patients may receive combination chemotherapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, mercaptopurine, cytarabine, thioguanine) by infusion, injection, intrathecally, and by mouth for up to 8 weeks.
- Prenisone, Capezzi Methotrexate (Down's Syndrome): Patients in regimen PC will receive cytarabine, vincristine sulfate, daunorubicin hydrochloride, and pegaspargase. They will also receive prednisone by mouth or infusion twice a day in weeks 1-4 and intrathecal methotrexate in weeks 2 and 5. Some patients in all groups may receive induction therapy for 2 additional weeks. Beginning in week 6 or 7, patients may receive combination chemotherapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, mercaptopurine, cytarabine, thioguanine) by infusion, injection, intrathecally, and by mouth for up to 8 weeks.
Arm/Group | Dexamethasone and Capizzi Methotrexate Patients < 10 Years | Dexamethasone, High Dose Methotrexate (Non Randomly Assigned) | Dexamethasone & Capizzi Methotrexate Patients => 10 Years Old | Dexamethasone, High Dose Methotrexate (IM) < 10 Years | Prednisone, Capizzi Methotrexate <10 Years | Prednisone, Capezzi Methotrexate >= 10 Years | Predisone and High Dose Methotrexate < 10 Yrs Old | Prenisone and High Dose Methotrexate >=10 Years | Dexamethasone, High Dose Methotrexate (IM) >= 10 Years | Prenisone, Capezzi Methotrexate (Down's Syndrome) | Dexamethasone, Capizzi Methotrexate Down Syndrome (Non Random)
Number analyzed (Participants) | 218 | 90 | 261 | 206 | 214 | 598 | 213 | 601 | 262 | 30 | 9
percentage of participants | 83.2 [76.6 to 89.9] | 81.6 [71.2 to 91.9] | 69.1 [63.1 to 75.2] | 91.2 [85.7 to 96.7] | 82.1 [75.3 to 89.0] | 73.5 [67.4 to 79.7] | 80.8 [73.6 to 88.0] | 75.8 [70.0 to 81.6] | 77.0 [71.5 to 82.6] | 61.8 [43.1 to 80.5] | 44.4 [12.0 to 76.9]

2. Secondary Outcome: Correlation of Minimal Residual Disease (MRD) Positive With Overall Survival (OS)
Description: Bone marrow MRD status is defined as positive with >= 0.1 detectable leukemia cells, and negative with < 0.1 detectable leukemia cells.
Time Frame: 5 Years
Population: Groups "Prednisone Capizzi MTX (Down's Syndrome)", "Dexamethasone, Capizzi MTX (non-random)" & "Prednisone and High Dose MTX (non-random) are not included in this OM as no patients survived the 5 year window for analysis. Cohort of MRD Positive patients who either had EFS/OS events occur before 5 years or did not have minimum 5 years of follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Prednisone, Capizzi Methotrexate >= 10 Years: Patients in regimen PC will receive cytarabine, vincristine sulfate, daunorubicin hydrochloride, and pegaspargase. They will also receive prednisone by mouth or infusion twice a day in weeks 1-4 and intrathecal methotrexate in weeks 2 and 5. Some patients in all groups may receive induction therapy for 2 additional weeks. Beginning in week 6 or 7, patients may receive combination chemotherapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, mercaptopurine, cytarabine, thioguanine) by infusion, injection, intrathecally, and by mouth for up to 8 weeks.
Arm/Group | Dexamethasone and Capizzi Methotrexate Patients < 10 Years | Dexamethasone, High Dose Methotrexate (Non Randomly Assigned) | Dexamethasone & Capizzi Methotrexate Patients => 10 Years Old | Dexamethasone, High Dose Methotrexate (IM) < 10 Years | Prednisone, Capizzi Methotrexate <10 Years | Prednisone, Capizzi Methotrexate >= 10 Years | Predisone and High Dose Methotrexate < 10 Yrs Old | Prednisone and High Dose Methotrexate >=10 Years | Dexamethasone, High Dose Methotrexate (IM) >= 10 Years
Number analyzed (Participants) | 28 | 13 | 53 | 15 | 17 | 116 | 20 | 112 | 44
percentage of participants | 79.2 [59.5 to 98.8] | 69.9 [32.4 to 100] | 65.6 [50.2 to 81.0] | 86.2 [49.9 to 100] | 93.8 [70.8 to 100] | 63.1 [49.4 to 76.8] | 84.2 [66.53 to 100] | 73.6 [59.8 to 87.4] | 74.6 [60.9 to 88.3]

3. Secondary Outcome: Correlation of Minimal Residual Disease (MRD) Negative With Overall Survival (OS).
Description: Bone marrow MRD status is defined as negative with < .01 detectable leukemia cells.
Time Frame: 5 years
Population: Patients on Arm/Group "Prednisone and High Dose Methotrexate (non randomly assigned)" are not included in the OM as there were no survivors for the 5 year duration. Cohort of MRD Negative patients some of whom have had EFS/OS events after 5 years or have minimum 5 years of follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Prednisone, Capizzi Methotrexate (Down's Syndrome): Patients in regimen PC will receive cytarabine, vincristine sulfate, daunorubicin hydrochloride, and pegaspargase. They will also receive prednisone by mouth or infusion twice a day in weeks 1-4 and intrathecal methotrexate in weeks 2 and 5. Some patients in all groups may receive induction therapy for 2 additional weeks. Beginning in week 6 or 7, patients may receive combination chemotherapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, mercaptopurine, cytarabine, thioguanine) by infusion, injection, intrathecally, and by mouth for up to 8 weeks.
Arm/Group | Dexamethasone and Capizzi Methotrexate Patients < 10 Years | Dexamethasone, High Dose Methotrexate (Non Randomly Assigned) | Dexamethasone & Capizzi Methotrexate Patients => 10 Years Old | Dexamethasone, High Dose Methotrexate (IM) < 10 Years | Prednisone, Capizzi Methotrexate <10 Years | Prednisone, Capizzi Methotrexate >= 10 Years | Prednisone and High Dose Methotrexate < 10 Yrs Old | Prednisone and High Dose Methotrexate >=10 Years | Dexamethasone, High Dose Methotrexate (IM) >= 10 Years | Prednisone, Capizzi Methotrexate (Down's Syndrome) | Dexamethasone, Capizzi Methotrexate Down Syndrome (Non Random)
Number analyzed (Participants) | 185 | 73 | 198 | 189 | 195 | 472 | 191 | 480 | 209 | 25 | 4
percentage of participants | 95.4 [91.3 to 99.4] | 92.9 [85.4 to 100] | 87.4 [82.5 to 92.4] | 98.1 [95.4 to 100] | 93.3 [88.6 to 98.0] | 90.2 [85.5 to 94.9] | 94.5 [90.0 to 98.9] | 90.5 [86.1 to 95.0] | 91.6 [87.5 to 95.8] | 78.3 [61.0 to 95.7] | 25.0 [-17.4 to 67.4]

4. Secondary Outcome: Correlation of Early Marrow Response Status With MRD Positive.
Description: Bone marrow status is defined as: M1: < 5% lymphoblasts; M2: 5-25% lymphoblasts; M3: > 25% lymphoblasts. Bone marrow MRD status is defined as positive with >= 0.1 detectable leukemia cells, and negative with < 0.1 detectable leukemia cells.
Time Frame: Day 29
Measure: Number; unit: participants
Arm/Group | Dexamethasone and Capizzi Methotrexate Patients < 10 Years | Dexamethasone, High Dose Methotrexate (Non Randomly Assigned) | Dexamethasone & Capizzi Methotrexate Patients => 10 Years Old | Dexamethasone, High Dose Methotrexate (IM) < 10 Years | Prednisone, Capizzi Methotrexate <10 Years | Prednisone, Capezzi Methotrexate >= 10 Years | Prednisone and High Dose Methotrexate < 10 Yrs Old | Prednisone and High Dose Methotrexate >=10 Years | Dexamethasone, High Dose Methotrexate (IM) >= 10 Years | Prednisone, Capezzi Methotrexate (Down's Syndrome) | Dexamethasone, Capizzi Methotrexate Down Syndrome (Non Random) | Prednisone and High Dose Methotrexate (Non Randomly Assigned)
Number analyzed (Participants) | 28 | 13 | 53 | 15 | 17 | 116 | 20 | 112 | 44 | 3 | 3 | 5
participants | 26 | 12 | 43 | 14 | 16 | 95 | 17 | 98 | 39 | 3 | 3 | 3

5. Secondary Outcome: Correlation of Early Marrow Response Status With MRD Negative.
Description: as for outcome 4
Time Frame: Day 29
Measure: Number; unit: participants
Arm/Group | Dexamethasone and Capizzi Methotrexate Patients < 10 Years | Dexamethasone, High Dose Methotrexate (Non Randomly Assigned) | Dexamethasone & Capizzi Methotrexate Patients => 10 Years Old | Dexamethasone, High Dose Methotrexate (IM) < 10 Years | Prednisone, Capizzi Methotrexate <10 Years | Prednisone, Capezzi Methotrexate >= 10 Years | Prednisone and High Dose Methotrexate < 10 Yrs Old | Prednisone and High Dose Methotrexate >=10 Years | Dexamethasone, High Dose Methotrexate (IM) >= 10 Years | Prednisone, Capezzi Methotrexate (Down's Syndrome) | Dexamethasone, Capizzi Methotrexate Down Syndrome (Non Random) | Prednisone and High Dose Methotrexate (Non Randomly Assigned)
Number analyzed (Participants) | 185 | 73 | 198 | 189 | 195 | 472 | 191 | 480 | 209 | 25 | 4 | 18
participants | 182 | 72 | 198 | 188 | 195 | 471 | 190 | 479 | 208 | 25 | 3 | 18

6. Secondary Outcome: Correlation of Minimal Residual Disease (MRD) Positive With Event Free Survival (EFS)
Description: Bone marrow MRD status is defined as positive with >= 0.1 detectable leukemia cells.
Time Frame: 5 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dexamethasone and Capizzi Methotrexate Patients < 10 Years | Dexamethasone, High Dose Methotrexate (Non Randomly Assigned) | Dexamethasone & Capizzi Methotrexate Patients => 10 Years Old | Dexamethasone, High Dose Methotrexate (IM) < 10 Years | Prednisone, Capizzi Methotrexate <10 Years | Prednisone, Capizzi Methotrexate >= 10 Years | Prednisone and High Dose Methotrexate < 10 Yrs Old | Prednisone and High Dose Methotrexate >=10 Years | Dexamethasone, High Dose Methotrexate (IM) >= 10 Years
Number analyzed (Participants) | 28 | 13 | 53 | 15 | 17 | 116 | 20 | 112 | 44
percentage of participants | 66.5 [43.7 to 89.2] | 43.3 [6.4 to 80.2] | 35.4 [21.4 to 49.3] | 80 [30.4 to 100] | 34.7 [-4.2 to 73.5] | 39 [25.7 to 52.4] | 55 [29.4 to 80.6] | 47.8 [32.3 to 63.3] | 49.4 [34.0 to 64.8]

7. Secondary Outcome: Correlation of Minimal Residual Disease (MRD) Negative With Event Free Survival (EFS).
Description: Bone marrow MRD status is defined as negative with < 0.1 detectable leukemia cells.
Time Frame: 5 years
Population: Group "Prednisone and High Dose MTX (non-random)" who either had EFS/OS events occur before 5 years or did not have minimum 5 years of follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dexamethasone and Capizzi Methotrexate Patients < 10 Years | Dexamethasone, High Dose Methotrexate (Non Randomly Assigned) | Dexamethasone & Capizzi Methotrexate Patients => 10 Years Old | Dexamethasone, High Dose Methotrexate (IM) < 10 Years | Prednisone, Capizzi Methotrexate <10 Years | Prednisone, Capezzi Methotrexate >= 10 Years | Prednisone and High Dose Methotrexate < 10 Yrs Old | Prednisone and High Dose Methotrexate >=10 Years | Dexamethasone, High Dose Methotrexate (IM) >= 10 Years | Prednisone, Capezzi Methotrexate (Down's Syndrome) | Dexamethasone, Capizzi Methotrexate Down Syndrome (Non Random)
Number analyzed (Participants) | 185 | 73 | 198 | 189 | 195 | 472 | 191 | 480 | 209 | 25 | 4
percentage of participants | 86.4 [79.8 to 93.1] | 93.6 [86.3 to 100] | 80.5 [74.5 to 86.4] | 93.1 [88.1 to 98.2] | 86.5 [80.2 to 92.8] | 83.4 [77.5 to 89.4] | 84.2 [77.2 to 91.3] | 83.9 [78.3 to 89.5] | 85.3 [80. to 90.5] | 74.4 [55.9 to 92.8] | 25 [-17.4 to 67.4]

ADVERSE EVENTS:
Description: SAE field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs.
Arm/Group | Dexamethasone and Capizzi Methotrexate Patients < 10 Years | Dexamethasone, High Dose Methotrexate (Non Randomly Assigned) | Dexamethasone & Capizzi Methotrexate Patients => 10 Years Old | Dexamethasone, High Dose Methotrexate (IM) < 10 Years | Prednisone, Capizzi Methotrexate <10 Years | Prednisone, Capezzi Methotrexate >= 10 Years | Prednisone and High Dose Methotrexate < 10 Yrs Old | Prednisone and High Dose Methotrexate >=10 Years | Dexamethasone, High Dose Methotrexate (IM) >= 10 Years | Prednisone, Capezzi Methotrexate (Down's Syndrome) | Dexamethasone, Capizzi Methotrexate Down Syndrome (Non Random) | Prednisone and High Dose Methotrexate (Non Randomly Assigned)
Serious Adverse Events (participants affected / at risk) | 16/218 | 17/90 | 42/261 | 25/206 | 20/214 | 64/598 | 16/213 | 67/601 | 27/262 | 3/30 | 3/9 | 1/23
Other Adverse Events (participants affected / at risk) | 215/218 | 87/90 | 250/261 | 203/206 | 212/214 | 564/598 | 204/213 | 576/601 | 256/262 | 30/30 | 9/9 | 20/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone and Capizzi Methotrexate Patients < 10 Years (N=218) | Dexamethasone, High Dose Methotrexate (Non Randomly Assigned) (N=90) | Dexamethasone & Capizzi Methotrexate Patients => 10 Years Old (N=261) | Dexamethasone, High Dose Methotrexate (IM) < 10 Years (N=206) | Prednisone, Capizzi Methotrexate <10 Years (N=214) | Prednisone, Capezzi Methotrexate >= 10 Years (N=598) | Prednisone and High Dose Methotrexate < 10 Yrs Old (N=213) | Prednisone and High Dose Methotrexate >=10 Years (N=601) | Dexamethasone, High Dose Methotrexate (IM) >= 10 Years (N=262) | Prednisone, Capezzi Methotrexate (Down's Syndrome) (N=30) | Dexamethasone, Capizzi Methotrexate Down Syndrome (Non Random) (N=9) | Prednisone and High Dose Methotrexate (Non Randomly Assigned) (N=23)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 6 (6) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (5) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 4 (5) | 0 (0) | 4 (4) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 6 (7) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (7) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GGT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 3 (7) | 6 (6) | 11 (13) | 2 (2) | 2 (2) | 13 (17) | 4 (4) | 12 (17) | 5 (8) | 1 (1) | 2 (2) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (1) | 5 (5) | 6 (6) | 3 (3) | 5 (6) | 4 (4) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 1 (2) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pregnancy, puerperium and perinatal conditions - Other, specify (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vagus nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone and Capizzi Methotrexate Patients < 10 Years (N=218) | Dexamethasone, High Dose Methotrexate (Non Randomly Assigned) (N=90) | Dexamethasone & Capizzi Methotrexate Patients => 10 Years Old (N=261) | Dexamethasone, High Dose Methotrexate (IM) < 10 Years (N=206) | Prednisone, Capizzi Methotrexate <10 Years (N=214) | Prednisone, Capezzi Methotrexate >= 10 Years (N=598) | Prednisone and High Dose Methotrexate < 10 Yrs Old (N=213) | Prednisone and High Dose Methotrexate >=10 Years (N=601) | Dexamethasone, High Dose Methotrexate (IM) >= 10 Years (N=262) | Prednisone, Capezzi Methotrexate (Down's Syndrome) (N=30) | Dexamethasone, Capizzi Methotrexate Down Syndrome (Non Random) (N=9) | Prednisone and High Dose Methotrexate (Non Randomly Assigned) (N=23)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 6 (6) | 2 (2) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 12 (13) | 12 (15) | 38 (45) | 16 (20) | 12 (13) | 52 (68) | 9 (9) | 35 (46) | 16 (23) | 1 (1) | 1 (1) | 1 (1)
Accessory nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 5 (7) | 3 (4) | 4 (4) | 1 (1) | 3 (3) | 10 (10) | 0 (0) | 14 (14) | 6 (7) | 2 (2) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 4 (5) | 5 (6) | 11 (18) | 6 (8) | 4 (5) | 18 (19) | 6 (6) | 18 (22) | 10 (13) | 2 (2) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 12 (13) | 1 (1) | 2 (2) | 16 (17) | 1 (1) | 13 (13) | 12 (15) | 1 (1) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 4 (5) | 7 (8) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 6 (8) | 3 (3) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 96 (272) | 33 (88) | 122 (305) | 94 (294) | 92 (263) | 274 (780) | 101 (352) | 275 (749) | 125 (303) | 12 (27) | 2 (3) | 10 (18)
Alcohol intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 3 (4) | 4 (5) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 2 (2)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (2) | 2 (2) | 9 (9) | 1 (2) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 30 (33) | 9 (9) | 36 (40) | 29 (29) | 24 (24) | 97 (106) | 24 (25) | 83 (86) | 38 (40) | 0 (0) | 0 (0) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 71 (147) | 33 (71) | 70 (128) | 68 (134) | 63 (123) | 179 (317) | 68 (122) | 167 (280) | 88 (169) | 13 (27) | 4 (5) | 5 (8)
Anorectal infection (Infections and infestations) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 16 (21) | 17 (19) | 43 (68) | 21 (30) | 18 (32) | 51 (68) | 15 (21) | 38 (53) | 20 (24) | 4 (4) | 4 (4) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (4) | 7 (8) | 2 (3) | 0 (0) | 4 (4) | 0 (0) | 12 (16) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arachnoiditis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (13) | 12 (14) | 2 (2) | 1 (1) | 22 (22) | 1 (1) | 17 (19) | 11 (13) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 6 (6) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 44 (66) | 22 (35) | 63 (91) | 54 (78) | 42 (60) | 146 (257) | 54 (97) | 143 (202) | 71 (121) | 5 (7) | 1 (1) | 4 (6)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asystole (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 1 (1) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (20) | 19 (22) | 1 (1) | 3 (7) | 26 (35) | 1 (1) | 35 (53) | 22 (33) | 1 (2) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 18 (19) | 1 (1) | 3 (3) | 44 (51) | 3 (3) | 34 (39) | 20 (23) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 7 (7) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3 (7) | 1 (1) | 3 (3) | 3 (3) | 7 (9) | 5 (5) | 4 (8) | 6 (6) | 3 (5) | 2 (2) | 0 (0) | 0 (0)
Blood antidiuretic hormone abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 15 (17) | 13 (17) | 47 (83) | 15 (18) | 4 (4) | 104 (178) | 7 (9) | 95 (133) | 50 (74) | 2 (2) | 2 (3) | 2 (2)
Blood corticotrophin decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 10 (11) | 0 (0) | 1 (1) | 11 (14) | 1 (1) | 14 (15) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 2 (3) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 11 (11) | 5 (5) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 16 (25) | 10 (19) | 9 (9) | 10 (12) | 10 (14) | 29 (37) | 24 (30) | 23 (25) | 8 (9) | 3 (5) | 1 (1) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 7 (8) | 0 (0) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 4 (8) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 6 (7) | 2 (3) | 9 (9) | 6 (6) | 2 (2) | 9 (9) | 1 (1) | 7 (10) | 3 (4) | 2 (2) | 1 (1) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1 (2) | 4 (5) | 1 (1) | 8 (9) | 6 (6) | 17 (20) | 7 (7) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 4 (4) | 3 (3) | 3 (4) | 7 (7) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 9 (11) | 2 (2) | 1 (1) | 7 (7) | 0 (0) | 9 (9) | 7 (8) | 1 (1) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 9 (12) | 13 (21) | 34 (41) | 21 (27) | 17 (19) | 73 (85) | 20 (22) | 59 (71) | 30 (37) | 5 (6) | 3 (3) | 3 (3)
Delayed puberty (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 8 (8) | 0 (0) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 15 (23) | 2 (2) | 1 (3) | 15 (16) | 0 (0) | 10 (14) | 7 (8) | 0 (0) | 0 (0) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 18 (22) | 7 (7) | 20 (24) | 24 (33) | 18 (22) | 35 (39) | 16 (19) | 36 (39) | 17 (21) | 7 (7) | 3 (3) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 7 (8) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 6 (7) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4) | 1 (1) | 1 (1) | 7 (8) | 1 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1) | 2 (2) | 4 (4) | 1 (2) | 1 (1) | 15 (15) | 2 (7) | 18 (19) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 11 (12) | 1 (1) | 0 (0) | 7 (8) | 1 (1) | 8 (8) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitis infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalomyelitis infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 4 (5) | 7 (7) | 1 (1) | 3 (3) | 16 (16) | 1 (1) | 14 (15) | 7 (7) | 0 (0) | 0 (0) | 3 (3)
Endocarditis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 3 (4) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 9 (12) | 5 (8) | 17 (19) | 14 (16) | 8 (10) | 24 (29) | 13 (14) | 16 (17) | 10 (10) | 3 (3) | 2 (5) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 12 (12) | 2 (4) | 2 (2) | 10 (10) | 3 (3) | 11 (11) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 3 (3) | 9 (9) | 2 (2) | 1 (1) | 15 (18) | 1 (1) | 11 (11) | 9 (10) | 0 (0) | 0 (0) | 0 (0)
Euphoria (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 4 (5) | 7 (9) | 3 (3) | 5 (5) | 13 (17) | 2 (2) | 17 (18) | 6 (6) | 0 (0) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 164 (387) | 52 (124) | 141 (279) | 134 (318) | 140 (314) | 278 (504) | 140 (318) | 283 (514) | 139 (268) | 22 (49) | 4 (6) | 12 (16)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 26 (34) | 3 (4) | 16 (17) | 15 (19) | 20 (26) | 26 (36) | 19 (23) | 27 (34) | 9 (10) | 3 (3) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 7 (12) | 7 (8) | 20 (22) | 8 (11) | 9 (12) | 41 (53) | 10 (15) | 32 (37) | 15 (16) | 3 (4) | 1 (1) | 2 (2)
Flashing lights (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (6) | 2 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 15 (15) | 2 (2) | 7 (7) | 6 (7) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5 (5) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 6 (6) | 1 (1) | 4 (7) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (3) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 6 (6) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GGT increased (Investigations) | 5 (10) | 6 (7) | 10 (16) | 5 (10) | 7 (12) | 36 (75) | 8 (14) | 35 (58) | 10 (12) | 1 (1) | 1 (1) | 1 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Glossopharyngeal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 6 (9) | 8 (9) | 0 (0) | 1 (1) | 17 (20) | 0 (0) | 22 (24) | 11 (11) | 0 (0) | 0 (0) | 1 (1)
Gum infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 11 (17) | 34 (45) | 2 (2) | 2 (3) | 81 (115) | 4 (4) | 74 (104) | 31 (40) | 2 (3) | 0 (0) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Hepatic hemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Hepatic necrosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 6 (8) | 0 (0) | 8 (9) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 6 (6) | 2 (2) | 0 (0) | 6 (7) | 0 (0) | 4 (4) | 6 (8) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 28 (28) | 20 (33) | 84 (126) | 24 (26) | 21 (23) | 155 (214) | 20 (25) | 159 (222) | 86 (131) | 14 (29) | 6 (9) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5) | 8 (8) | 13 (13) | 4 (5) | 5 (5) | 23 (28) | 6 (6) | 19 (19) | 10 (11) | 6 (7) | 1 (2) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 8 (8) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 7 (7) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 4 (4) | 1 (1) | 2 (2) | 6 (6) | 0 (0) | 4 (4) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 7 (7) | 3 (3) | 10 (17) | 4 (4) | 6 (7) | 16 (17) | 10 (10) | 15 (16) | 8 (11) | 0 (0) | 1 (1) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 4 (6) | 10 (14) | 0 (0) | 5 (6) | 13 (16) | 0 (0) | 13 (18) | 10 (12) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 3 (4) | 2 (2) | 2 (2) | 11 (12) | 1 (1) | 7 (7) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 19 (25) | 10 (12) | 24 (33) | 11 (14) | 8 (9) | 37 (45) | 6 (6) | 28 (32) | 16 (19) | 5 (11) | 3 (4) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 21 (23) | 14 (15) | 26 (31) | 15 (20) | 11 (12) | 56 (58) | 5 (5) | 51 (54) | 32 (38) | 6 (7) | 4 (6) | 2 (2)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 8 (10) | 3 (3) | 4 (4) | 7 (7) | 13 (14) | 6 (9) | 8 (9) | 7 (9) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 30 (43) | 33 (60) | 49 (68) | 42 (60) | 30 (39) | 98 (127) | 48 (69) | 126 (170) | 59 (78) | 6 (8) | 4 (5) | 6 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 4 (5) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 34 (36) | 22 (27) | 46 (54) | 26 (31) | 20 (23) | 84 (100) | 19 (21) | 78 (89) | 51 (63) | 5 (6) | 4 (5) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (6) | 8 (9) | 15 (20) | 6 (6) | 2 (2) | 34 (36) | 6 (6) | 15 (18) | 13 (13) | 1 (1) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 5 (6) | 6 (6) | 16 (16) | 6 (6) | 4 (5) | 30 (33) | 3 (3) | 22 (23) | 16 (16) | 2 (2) | 2 (2) | 2 (2)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 14 (14) | 20 (26) | 10 (12) | 9 (10) | 34 (40) | 8 (8) | 32 (33) | 12 (14) | 5 (6) | 4 (5) | 0 (0)
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 5 (5) | 8 (8) | 4 (4) | 1 (1) | 8 (8) | 3 (3) | 7 (13) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 147 (347) | 63 (179) | 149 (322) | 141 (347) | 146 (324) | 297 (595) | 136 (322) | 288 (545) | 145 (290) | 23 (76) | 7 (25) | 14 (27)
Infective myositis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1) | 6 (10) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 5 (5) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (3) | 3 (4) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Intraoperative respiratory injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraoperative skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 19 (26) | 3 (6) | 12 (16) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 4 (11) | 1 (1) | 3 (4) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Joint infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 8 (8) | 7 (8) | 39 (69) | 10 (12) | 10 (14) | 44 (58) | 6 (8) | 35 (52) | 12 (17) | 1 (1) | 1 (1) | 3 (3)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 29 (37) | 5 (5) | 21 (23) | 14 (16) | 17 (21) | 40 (47) | 19 (23) | 47 (52) | 10 (11) | 3 (6) | 1 (1) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 15 (38) | 9 (29) | 14 (32) | 21 (48) | 16 (32) | 35 (73) | 17 (33) | 38 (93) | 10 (23) | 2 (3) | 1 (1) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 2 (2) | 1 (2) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 22 (28) | 19 (24) | 57 (63) | 27 (32) | 13 (13) | 134 (155) | 31 (38) | 99 (113) | 48 (61) | 11 (14) | 4 (5) | 3 (3)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 7 (8) | 2 (2) | 6 (9) | 5 (11) | 1 (1) | 1 (1) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Myelitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (8) | 5 (7) | 26 (29) | 7 (9) | 2 (2) | 64 (86) | 4 (4) | 48 (60) | 32 (39) | 4 (4) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (3) | 1 (1) | 7 (7) | 2 (2) | 0 (0) | 12 (12) | 2 (3) | 13 (15) | 6 (6) | 1 (2) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 2 (2) | 0 (0) | 4 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 184 (682) | 61 (248) | 187 (585) | 168 (636) | 172 (595) | 437 (1393) | 168 (652) | 442 (1279) | 188 (661) | 23 (85) | 7 (13) | 15 (42)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 8 (9) | 0 (0) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 4 (17) | 4 (11) | 0 (0) | 0 (0) | 0 (0)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 5 (5) | 11 (12) | 3 (3) | 7 (8) | 23 (24) | 9 (10) | 12 (13) | 8 (8) | 2 (2) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 16 (18) | 3 (3) | 1 (1) | 9 (9) | 13 (15) | 5 (5) | 12 (12) | 8 (8) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 6 (7) | 10 (11) | 4 (4) | 3 (3) | 25 (31) | 3 (3) | 30 (31) | 7 (8) | 1 (1) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (7) | 13 (15) | 2 (2) | 8 (8) | 22 (24) | 4 (4) | 27 (33) | 17 (19) | 1 (1) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreas infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (4) | 5 (6) | 16 (21) | 6 (7) | 4 (6) | 31 (34) | 5 (5) | 16 (26) | 7 (7) | 1 (1) | 0 (0) | 1 (1)
Papilledema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Penile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 12 (21) | 12 (14) | 34 (67) | 10 (20) | 13 (18) | 68 (100) | 6 (16) | 54 (97) | 31 (60) | 5 (9) | 1 (1) | 5 (8)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (20) | 7 (10) | 22 (27) | 8 (10) | 4 (4) | 42 (64) | 9 (18) | 37 (62) | 15 (19) | 1 (2) | 0 (0) | 3 (4)
Peritoneal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 1 (1) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 7 (7) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (4) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 7 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Phlebitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 96 (199) | 39 (85) | 101 (217) | 78 (151) | 77 (130) | 249 (481) | 74 (125) | 226 (444) | 102 (223) | 16 (31) | 5 (8) | 8 (12)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 5 (5) | 5 (5) | 1 (1) | 13 (15) | 3 (3) | 8 (8) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5) | 9 (9) | 6 (7) | 6 (7) | 13 (13) | 5 (7) | 11 (11) | 10 (11) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 7 (9) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyramidal tract syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 7 (7) | 7 (8) | 4 (4) | 6 (6) | 1 (1) | 4 (5) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (3) | 5 (11) | 3 (4) | 8 (8) | 3 (3) | 6 (7) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 3 (3) | 9 (10) | 4 (4) | 3 (4) | 19 (21) | 5 (5) | 15 (18) | 5 (5) | 2 (2) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 3 (5) | 1 (1) | 3 (3) | 4 (4) | 17 (21) | 3 (3) | 12 (13) | 2 (3) | 2 (3) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 4 (4) | 4 (5) | 17 (32) | 10 (11) | 6 (6) | 25 (31) | 5 (7) | 22 (26) | 8 (10) | 0 (0) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 6 (6) | 6 (10) | 9 (10) | 7 (9) | 5 (5) | 15 (17) | 6 (10) | 11 (13) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 5 (6) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 9 (11) | 8 (9) | 13 (14) | 6 (6) | 15 (15) | 40 (44) | 8 (9) | 32 (34) | 9 (10) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestine infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 5 (6) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Soft tissue necrosis upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spleen disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (3) | 7 (8) | 0 (0) | 1 (1) | 17 (19) | 3 (3) | 14 (15) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 8 (9) | 3 (4) | 3 (5) | 17 (21) | 2 (2) | 23 (26) | 13 (14) | 3 (4) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 8 (8) | 4 (4) | 3 (3) | 14 (14) | 1 (1) | 12 (12) | 11 (11) | 2 (2) | 0 (0) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 5 (5) | 5 (5) | 10 (11) | 7 (7) | 1 (1) | 13 (15) | 3 (3) | 12 (12) | 6 (6) | 0 (0) | 1 (1) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 28 (38) | 5 (8) | 14 (15) | 18 (24) | 21 (26) | 19 (20) | 17 (21) | 23 (26) | 9 (9) | 1 (1) | 0 (0) | 3 (3)
Urethral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (8) | 5 (7) | 8 (9) | 9 (11) | 11 (11) | 19 (22) | 7 (10) | 18 (18) | 9 (12) | 2 (2) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 2 (2) | 10 (10) | 1 (1) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vagus nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 4 (5) | 6 (6) | 0 (0) | 0 (0) | 12 (12) | 1 (1) | 11 (12) | 5 (6) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 1 (2) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 16 (16) | 11 (13) | 40 (47) | 16 (17) | 13 (17) | 78 (99) | 18 (20) | 74 (89) | 30 (36) | 5 (5) | 3 (3) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 4 (7) | 5 (19) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 11 (13) | 3 (3) | 17 (19) | 5 (15) | 4 (5) | 34 (44) | 8 (13) | 21 (24) | 12 (17) | 2 (2) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 91 (292) | 41 (125) | 103 (307) | 92 (289) | 83 (260) | 213 (603) | 81 (225) | 218 (549) | 124 (350) | 16 (46) | 5 (8) | 6 (15)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 2 (3) | 16 (17) | 3 (3) | 8 (10) | 4 (4) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The COG SDC reviewed the NLM notification related to ct.gov AE/SAE reporting. The information in 'Additional Description' is accurate with respect to data supplied to ct.gov.COG plans to submit data AE/SAE data consistent with the text in this field.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval